CLINICAL TRIAL: NCT00344149
Title: Rituximab as Second Line Treatment for ITP; A Multicenter, Randomized, Double Blind, Placebo-controlled, Phase III Study. "The RITP Study"
Brief Title: Rituximab as Second Line Treatment for ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); South-Eastern Regional Health Authority (Unknown)
Responsible Party: Principal Investigator, Waleed Ghanima, Dr Waleed Ghanima, MD. PhD, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3114; ITP001
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: Idiopathic Thrombocytopenic Purpura; Rituximab; Splenectomy; Response; Treatment; treatment of Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): I.V infusion of Rituximab 375 mg/m2 per week for 4 weeks
  Interventions: Drug: Rituximab (Mabthera)
- Placebo (Placebo Comparator): I.V infusion of NaCl 0.9%
  Interventions: Drug: Rituximab (Mabthera)

INTERVENTIONS:
Drug: Rituximab (Mabthera) — I.V infusion of Rituximab 375 mg/m2 per week for 4 weeks

SUMMARY:
Immune thrombocytopenic purpura (ITP) is an autoimmune disorder characterized thrombocytopenia.

Splenectomy is the standard treatment for patients who fails the first-line treatment: corticosteroid. Rituximab, has recently emerged as a promising treatment for ITP. The aim of the study is to determine whether early treatment with Rituximab can result in durable remissions, and consequently, lead to the avoidance of splenectomy in a significant number of patients.

DETAILED DESCRIPTION:
ITP is an autoimmune disorder characterized by formation of autoantibodies against platelet antigens leading to premature platelet destruction and persistent thrombocytopenia often resulting in bleeding.

The goal of treatment is to raise the platelet count to a hemostatically safe level.

Treatment with corticosteroids rarely results in durable responses, and most of the patients will ultimately require a second-line treatment. Splenectomy results in a high rate of sustained remissions. However, the procedure is invasive and is associated with considerable short and long term morbidity and mortality. Rituximab, a chimeric anti-CD20 antibody with a B-cell depleting effect, has recently emerged as a promising treatment for ITP.

The study aims to determine whether early treatment with Rituximab can result in durable remissions, and consequently, avoidance of splenectomy in a clinical significant number of patients.

The main objective of this study is to assess the rate of treatment failure (splenectomy or meeting criteria for splenectomy after week 12) at 1.5-year in a prospective, randomized, placebo-controlled, double-blind, multi-centre

ELIGIBILITY:
Inclusion Criteria:

1. ITP with platelet count <30 x 109 /l after 2 weeks of treatment with prednisolon or during prednisolon tapering period i.e. from week three of prednisolon initiation. Patients with platelet count between 30 -50 are eligible if a higher platelet count is considered necessary, because of : concomitant medical illness predisposing to bleeding (hypertension, GI bleeding, bleeding diathesis, previous history of bleeding) concomitant medical condition requiring platelet blocking agents/ anticoagulation, persistent bleeding despite platelets > 30 x 109 /l, prior to surgery, or because of other patient related factors necessitating higher platelet count as occupation, hobby, psychological intolerability.
2. Subject is >18 years
3. Subject has signed and dated written informed consent.
4. Subject is able to understand and comply with protocol requirements and instructions, and intends to complete the study as planned.
5. Females in fertile age should express willingness for use of contraceptive means for 6 months following the administration of the study drugs.

Exclusion criteria:

1. Previous splenectomy, chemotherapy, treatment with anti-D Ig, rituximab, or immune-suppressive treatments other than corticosteroids, Dapsone or Danazol
2. Underlying malignancy or previous history of malignancy in the past 5 years (except skin carcinoma)
3. Pregnancy and lactation
4. Not willing to participate in the study
5. Expected survival of < 2 years
6. Known intolerance to murine antibodies
7. Females in child-bearing age not willing to use contraception for 6 months
8. HIV-positive/AIDS-, Hepatitis -B virus positive- or Hepatitis -C virus positive
9. Patients with a definite Systemic Lupus Erythematosus (SLE) (> 4 of the American College of Rheumatology Criteria)
10. Patients currently involved in another clinical trial with evaluation of drug treatment
11. Bacterial infections, viral infections, fungal infections, myco-bacterial infections (excluding fungal infections) or other evolutive infections or any other infections episode requiring hospitalisation or treatment with an antibiotics 4 weeks before selection for IV route or within 2 weeks before selection for oral route
12. History of soft tissue, bone or joint infections (fascitis, abscess, osteomyelitis, septic arthritis) during the last year prior to inclusion in the study
13. Medical history of relapsing or chronic severe infectious diseases or any other underlying pathology predisposing to serious infections
14. Known Primary or secondary immune deficiency syndromes
15. Administration of a living vaccine within 4 weeks preceding the inclusion in the study -16- Previous treatment with any lymphocytes depleting medication (e.g.: MabCampath®)

17- Previous treatment with inhibitors of leucocytes transmigration (e.g.: Tysabri®) 18- Known intolerance to human monoclonal antibodies 19- Known severe chronic pulmonary obstructive Disease (FEV < 50% or functional dyspnoea grade 3) 20- Known congestive heart failure NYHA (New York Heart Association classification of heart failure) class III and IV 21- Recent episode (<6 months) of acute coronary syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is treatment failure as defined by a composite end point of Splenectomy performed at any time after randomization or Meeting the predefined Criteria for Splenectomy at or after week 12 that is if splenectomy is not performed. | 1.5 years

SECONDARY OUTCOMES:
Response rates | 1.5 years
Relapse rate | 1.5 years
Mortality rate | 1.5 years
Complications rate | 1.5 years
  Including bleeding, infections and thromboembolic events

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghanima, MD, Principal Investigator — Østfold Hospital trust in Fredrikstad; Pål Andre Holme, Principal Investigator — Oslo University Hospital; Finn Wisløff, MD, PhD, Principal Investigator — Ullevaal University Hospital; Anders Waage, MD, PhD, Principal Investigator — St. Olavs Hospital, Trondheim, Norway; Geir Tjønnfjord, MD, PhD, Principal Investigator — Rikshospitalet- Oslo-Norway; Peter Meyer, MD, PhD, Principal Investigator — Rogaland sentralt sykehus - Stavanger-Norway; Marc Michel, MD, Principal Investigator — Dept. of Internal medicine Henri Mondor University Hospital Créteil- France
Locations (1):
- Østfold Hospital Trust in Fredrikstad and National hospital in Oslo, Fredrikstad and Oslo, Norway

REFERENCES:
- [Background] Cooper N, Stasi R, Cunningham-Rundles S, Feuerstein MA, Leonard JP, Amadori S, Bussel JB. The efficacy and safety of B-cell depletion with anti-CD20 monoclonal antibody in adults with chronic immune thrombocytopenic purpura. Br J Haematol. 2004 Apr;125(2):232-9. doi: 10.1111/j.1365-2141.2004.04889.x. PMID 15059147
- [Derived] Ghanima W, Khelif A, Waage A, Michel M, Tjonnfjord GE, Romdhan NB, Kahrs J, Darne B, Holme PA; RITP study group. Rituximab as second-line treatment for adult immune thrombocytopenia (the RITP trial): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2015 Apr 25;385(9978):1653-61. doi: 10.1016/S0140-6736(14)61495-1. Epub 2015 Feb 5. PMID 25662413